CLINICAL TRIAL: NCT04818957
Title: Vitamin D Replacement Using Oral Thin Film (OTF) Cholecalciferol in Patients Undergoing Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0151
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Vitamin D Deficiency; Hematopoietic Stem Cell Transplantation (HSCT)
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin D Oral Thin Film (OTF) (Experimental): Study subjects will receive vitamin D OTF for a maximum of 12 weeks.
  Interventions: Dietary Supplement: Oral Thin Film (OTF) Cholecalciferol (Vitamin D3)

INTERVENTIONS:
Dietary Supplement: Oral Thin Film (OTF) Cholecalciferol (Vitamin D3) — Study participants will receive vitamin D OTF weekly for a maximum of 12 weeks. The dose may be increased or decreased based on the dosing schema.

SUMMARY:
The investigators hypothesize that vitamin D levels can be improved in hematopoietic stem cell transplantation (HSCT) recipients not responding or tolerating standard enteral supplementation options by using vitamin D oral thin film (OTF) administration.

DETAILED DESCRIPTION:
The purpose of this study is to investigate efficacy of oral thin film (OTF) cholecalciferol (vitamin D3) replacement in hematopoietic stem cell transplantation (HSCT) recipients who failed to achieve or sustain adequate vitamin D levels after vitamin D supplementation using current standard of care, or those unable to take/tolerate currently available enteral vitamin D formulations. With oral thin film (OTF) cholecalciferol, investigators hope to significantly improve the ease of administration, restoring compliance and facilitating therapeutic vitamin D levels without relying on the gut for absorption.

ELIGIBILITY:
Inclusion Criteria:

* HSCT recipients of any age with vitamin D levels ≤35 ng/mL, or unable to tolerate, or refractory to enteral supplementation formulations of Vitamin D will be offered Vitamin D OTF.

Exclusion Criteria:

* Subjects with 25OHD level >60ng/mL. Subjects can be re-screened multiple times and enrolled later if they meet study criteria.
* Subjects with clinically significant and uncontrolled hypercalcemia as deemed by treating physician.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Vitamin D Level | 12 weeks from starting vitamin D supplementation
  Number of participants who achieve 25OH vitamin D level >35ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Allison Bartlett, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Gregory Wallace, DO, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bartlett AL, Zhang G, Wallace G, McLean S, Myers KC, Teusink-Cross A, Taggart C, Patel B, Davidson R, Davies SM, Jodele S. Optimized vitamin D repletion with oral thin film cholecalciferol in patients undergoing stem cell transplant. Blood Adv. 2023 Aug 22;7(16):4555-4562. doi: 10.1182/bloodadvances.2023009855. PMID 37285801